CLINICAL TRIAL: NCT06691984
Title: A Phase 3, Open-label, Multicenter, Randomized Study of Xaluritamig vs Cabazitaxel or Second Androgen Receptor-Directed Therapy in Subjects With Metastatic Castration-Resistant Prostate Cancer Previously Treated With Chemotherapy
Brief Title: Phase 3 Study of Xaluritamig vs Cabazitaxel or Second Androgen Receptor-Directed Therapy in Participants With Progressive Metastatic Castration-Resistant Prostate Cancer (XALute)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230005; 2024-513968-25 (Other: EU CTR Number)
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Oncology; Xaluritamig; Cabazitaxel; Prostate cancer; Abiraterone; Enzalutamide
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms | interventions — abiraterone; enzalutamide; cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Xaluritamig (Experimental): Participants with metastatic castration-resistant prostate cancer (mCRPC) will be randomized to receive Xaluritamig as an intravenous (IV) infusion.
  Interventions: Drug: Xaluritamig
- Cabazitaxel/Abiraterone/Enzalutamide (Active Comparator): Participants with mCRPC will be randomized to receive cabazitaxel as an IV infusion, or a second androgen receptor-directed therapy of either abiraterone as oral tablets, or enzalutamide as oral tablets at the investigator's discretion.
  Interventions: Drug: Abiraterone; Drug: Enzalutamide; Drug: Cabazitaxel

INTERVENTIONS:
Drug: Xaluritamig — Short-term IV infusion
  Arms: Xaluritamig
Drug: Abiraterone — Oral tablets
  Arms: Cabazitaxel/Abiraterone/Enzalutamide
Drug: Enzalutamide — Oral tablets
  Arms: Cabazitaxel/Abiraterone/Enzalutamide
Drug: Cabazitaxel — IV infusion
  Arms: Cabazitaxel/Abiraterone/Enzalutamide

SUMMARY:
The main objective of the study is to compare overall survival in participants receiving xaluritamig versus investigator's choice (cabazitaxel or second androgen receptor-directed therapy [ARDT]).

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent prior to initiation of any study-specific activities/procedures.
* Age ≥ 18 years (or ≥ legal age within the country if it is older than 18 years) at the time of signing the informed consent.
* Participant must have histological, pathological, and/or cytological confirmation of adenocarcinoma of the prostate. Mixed histologies (eg, adenocarcinoma with neuroendocrine component) are not permitted.
* mCRPC with ≥ 1 metastatic lesion that is present on baseline computed tomography (CT), magnetic resonance imaging (MRI), or bone scan imaging obtained within 28 days prior to enrollment.
* Evidence of progressive disease, defined as 1 or more PCWG3 criteria:

  * Serum PSA progression defined as 2 consecutive increases in PSA over a previous reference value measured at least 1 week prior. The minimal start value is 2.0 ng/mL.
  * Soft-tissue progression defined as an increase ≥ 20% in the sum of the diameter (SOD) (short axis for nodal lesions and long axis for non-nodal lesions) of all target lesions based on the smallest SOD since treatment started or the appearance of one or more new lesions or unequivocal progression of existing non-target lesions.
  * Progression of bone disease: defined by the appearance of at least 2 new bone lesion(s) by bone scan (as per the 2+2 PCWG3 criteria).
* Participants must have had a prior orchiectomy and/or ongoing androgen-deprivation therapy and a castrate level of serum testosterone (< 50 ng/dL or < 1.7 nmol/L).
* Prior progression on at least one ARDT (enzalutamide, abiraterone, apalutamide, darolutamide).
* Prior treatment with only one taxane therapy in the mCRPC setting. Note: Prior treatment with docetaxel in the metastatic hormone-sensitive prostate cancer (mHSPC) setting is permitted; however, participants must have also received one, and only one, taxane therapy in the mCRPC setting.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
* Adequate organ function.
* Life expectancy of ≥ 12 weeks per the treating physician's assessment.

Key Exclusion Criteria:

Prior & Concomitant Therapy:

* Prior six transmembrane epithelial antigen of the prostate 1 (STEAP1)-targeted therapy.
* Any anticancer therapy, immunotherapy, or investigational agent within 4 weeks prior to the first dose of study treatment, not including androgen receptor pathway inhibitors (ARPIs) (abiraterone, enzalutamide, darolutamide, apalutamide): minimum washout of 2 weeks prior to the first dose of study treatment and androgen suppression therapy (eg, luteinizing hormone-releasing hormone/gonadotropin-releasing hormone [LHRH/GnRH] analogue [agonist/antagonist]).
* Prior Prostate-Specific Membrane Antigen (PSMA) radioligand therapy (RLT) within 3 months of the first dose of study treatment unless participants received < 2 cycles of therapy.
* Prior palliative radiotherapy within 2 weeks of first dose of study treatment. Participants must have recovered from all radiation-related toxicities.
* Concurrent cytotoxic chemotherapy, ARDT, immunotherapy, radioligand therapy, PARP inhibitor, biological therapy, investigational therapy. Note: Prior treatment with a PARP inhibitor is permitted as long as not within 4 weeks before first dose of study treatment.
* Prior radionuclide therapy (Radium-223) within 2 months of first dose of study treatment.
* Treatment with live and live-attenuated vaccines within 4 weeks before the first dose of study treatment.

Disease Related:

* Participants with a history of central nervous system (CNS) metastasis. Note: Participants with treated, asymptomatic, and clinically stable dural metastases are eligible.
* Unresolved toxicities from prior anti-tumor therapy not having resolved to CTCAE version 5.0 events grade above 1 or baseline, with the exception of alopecia or toxicities that are stable and well controlled AND there is an agreement to allow inclusion by both the investigator and the sponsor.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2029-01-02 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 53 months

SECONDARY OUTCOMES:
Radiographic Progression-free Survival (rPFS) per Prostate Cancer Working Group 3 (PCWG3)-modified Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 53 months
Objective Response Rate per Modified RECIST v1.1 as Assessed by BICR | Up to approximately 53 months
Duration of Response (DOR) per Modified RECIST v1.1 as Assessed by BICR | Up to approximately 53 months
Disease Control Rate per Modified RECIST v1.1 as Assessed by BICR | Up to approximately 53 months
Time to Response (TTR) per Modified RECIST v1.1 as Assessed by BICR | Up to approximately 53 months
Time to First Symptomatic Skeletal Events (SSE) | Up to approximately 53 months
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to approximately 53 months
Change from Baseline in Brief Pain Inventory - Short Form (BPI-SF) Worst Pain Score | Baseline and approximately 53 months
Change from Baseline in BPI-SF Pain Intensity Scale Score | Baseline and approximately 53 months
Change from Baseline in BPI-SF Pain Interference Scale Score | Baseline and approximately 53 months
Change from baseline in the European Quality of Life 5 Domain 5 Level Scale (EQ-5D-5L) Utility Score | Baseline and approximately 53 months
Change from baseline in the EQ-5D-5L Visual Analogue Scale (VAS) | Baseline and approximately 53 months
Change from Baseline in Functional Assessment of Cancer Therapy - Prostate (FACT-P) Total Score and Subscale Score | Baseline and approximately 53 months
Time to Worsening in BPI-SF Worst Pain Score | Up to approximately 53 months
Time to Worsening in BPI-SF Pain Intensity Scale Score | Up to approximately 53 months
Time to Worsening in BPI-SF Pain Interference Scale Score | Up to approximately 53 months
Time to Worsening in FACT-P Total Score | Up to approximately 53 months
Time to Pain Improvement in Participants with Moderate/Severe Pain at Baseline | Up to approximately 53 months
Time to Pain Improvement after Worsening in BPI-SF Pain Intensity Scale Score | Up to approximately 53 months
Time to Pain Improvement after Worsening in BPI-SF Pain Interference Scale | Up to approximately 53 months
Number of Patient-Reported Symptomatic AEs per Patient-reported Outcome - Common Terminology Criteria for Adverse Events (PRO-CTCAE) Item Library | Up to approximately 53 months
Patient-Reported Summary Scores for Overall Bother of Side Effects per FACT-P | Up to approximately 53 months
Percentage of Participants Achieving a ≥50% Reduction in Prostate-specific Antigen (PSA) (PSA50) | Up to approximately 53 months
Percentage of Participants Achieving a ≥90% Reduction in PSA (PSA90) | Up to approximately 53 months
Maximum Serum Concentration (Cmax) of Xaluritamig | Up to approximately 53 months
Time to Cmax (Tmax) of Xaluritamig | Up to approximately 53 months
Minimum Serum Concentration (Cmin) of Xaluritamig | Up to approximately 53 months
Area Under the Concentration-time Curve (AUC) of Xaluritamig | Up to approximately 53 months
Accumulation Following Multiple Dosing of Xaluritamig | Up to approximately 53 months
Half-life (t1/2) of Xaluritamig | Up to approximately 53 months
Number of Participants with Anti-xaluritamig Antibody | Up to approximately 53 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (163):
- United States (42):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Providence Saint Jude Medical Center, Fullerton, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California Irvine, Orange, California
  - University of California San Francisco, San Francisco, California
  - University of Florida, College of Medicine, Gainesville, Florida
  - Sylvester Comprehensive Cancer Center-Fox Building, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Louisville Health - James Graham Brown Cancer Center, Louisville, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Henry Ford Health Systems, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Yale New Haven Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sanford Oncology Clinic and Pharmacy, Sioux Falls, South Dakota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - Virginia Oncology Associates, Norfolk, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - Macquarie University, North Ryde, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Medical Centre, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (7):
  - Medizinische Universitaet Graz, Graz
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Ordensklinikum Linz Elisabethinen, Linz
  - Landeskrankenhaus Salzburg, Salzburg
  - Universitaetsklinikum Sankt Poelten, Sankt Pölten
  - Krankenhaus der Barmherzigen Brueder Wien, Vienna
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
- Belgium (4):
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Algemeen Ziekenhuis Groeninge - Campus Kennedylaan, Kortrijk
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
- Canada (5):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - BC Cancer Vancouver, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sir Mortimer B Davis - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-Universite Laval, Québec, Quebec
- Denmark (2):
  - Aarhus University Hospital, Aarhus N
  - Vejle Sygehus, Vejle
- France (10):
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Saint Andre, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Grenoble - Hopital Nord Michallon, La Tronche
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Hopital d Instruction des Armees - Hopital Begin, Saint-Mandé
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - Gustave Roussy, Villejuif
- Germany (11):
  - Charite - Universitaetsmedizin Berlin, Campus Mitte, Berlin
  - Universitaetsklinikum Dresden, Dresden
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Schleswig-Holstein - Luebeck, Lübeck
  - Klinikum rechts der Isar der TUM, München
  - Universitaetsklinikum Muenster, Münster
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (5):
  - Alexandra Hospital, Athens
  - Athens Medical Center S.A - Iatriko Amarousiou, Athens
  - Metropolitan General, Athens
  - Metropolitan Hospital, Athens
  - European Interbalkan Medical Center, Thessaloniki
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong
- Italy (7):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Foggia, Foggia
  - Ospedale Sacro Cuore di Gesù Azienda Sanitaria Locale di Lecce, Gallipoli
  - Ospedale Policlinico San Martino IRCCS, Genova
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano
  - Ospedale Santa Chiara Azienda Provinciale per i Servizi Sanitari Provincia Autonoma di Trento, Trento
- Japan (15):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Gunma University Hospital, Maebashi, Gunma
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kitasato University Hospital, Sagamihara-shi, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Osaka International Cancer Institute, Osaka, Osaka
  - The University of Osaka Hospital, Suita-shi, Osaka
  - Saitama Medical University International Medical Center, Hidaka-shi, Saitama
  - Dokkyo Medical University Saitama Medical Center, Koshigaya-shi, Saitama
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - The Cancer institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
- Netherlands (5):
  - Nederlands Kanker Instituut Antoni van Leeuwenhoekziekenhuis, Amsterdam
  - Reinier de Graaf Gasthuis, Delft
  - Universitair Medisch Centrum Groningen, Groningen
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - SPZOZ Szpital Uniwersytecki w Krakowie, Krakow
- Singapore (3):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (6):
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (10):
  - Hospital Regional Universitario de Malaga, Málaga, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Instituto Valenciano de Oncologia, Valencia, Valencia
  - Institut Catala d Oncologia Hospitalet Hospital Duran i Reynals, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Sweden (4):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Skanes Universitetssjukhus, Lund
  - Karolinska Universitetssjukhuset, Stockholm
  - Norrlands Universitetssjukhus, Umeå
- Switzerland (5):
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Sankt Gallen, Sankt Gallen
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District
- Turkey (Türkiye) (3):
  - Ankara Universitesi Tip Fakultesi Hastanesi, Ankara
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul
  - Izmir Ekonomi Universitesi Medical Point Hastanesi, Izmir
- United Kingdom (5):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - University College London Hospital, London
  - Guys Hospital, London
  - Sarah Cannon Research Institute UK, London
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com